CLINICAL TRIAL: NCT02085083
Title: Improving OutcoMes in the Pediatric to Adult Care Transition in Inflammatory Bowel Disease
Acronym: IMPACT-IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IMPACT-IBD
Record Dates: First submitted 2013-12-23; First posted 2014-03-12 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Inflammatory Bowel Disease; Crohn Disease; Colitis, Ulcerative
Keywords: Inflammatory Bowel Disease; Transition; Adolescent; Chronic Disease; Colitis, Ulcerative
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular telephone and email access to an IBD Nurse (Experimental): The IBD pediatric-adult transition nurse will send an email to each individual randomized to the intervention arm each month. The email will include the following: Brief Questionnaire;The Option For Direct Nurse Contact; Educational modules; MyHealth Passport and a Comprehensive Study Questionnaire.
  Interventions: Behavioral: Telephone and email correspondence with an Inflammatory Bowel Disease Nurse
- Minimal Intervention (Active Comparator): The IBD pediatric-adult transition nurse will send an email to each individual randomized to the control arm every 3 months. The email will include the following: MyHealth Passport and Study Questionnaire. This intervention is not expected to significantly improve outcomes.
  Interventions: Behavioral: Minimal Intervention Arm

INTERVENTIONS:
Behavioral: Telephone and email correspondence with an Inflammatory Bowel Disease Nurse — The IBD pediatric-adult transition nurse will send an email each month containing:
  Brief Questionnaire: A link to a secured website will be provided where participants will respond to a questionnaire.
  Direct Nurse Contact: Telephone and email correspondence with an Inflammatory Bowel Disease Nurse
  Educational module: Every other month, we will include in the email another link to an optional educational module that will be part of a curriculum to facilitate transition readiness.
  MyHealth Passport
  Study Questionnaire: A personalized link to a more comprehensive study questionnaire similar to the baseline questionnaire will be emailed in the 6th and 12th (final) email.
  Arms: Regular telephone and email access to an IBD Nurse
Behavioral: Minimal Intervention Arm — Patients randomized to the control group will have receive email based questionnaires and information relating to the MyHealth Passport application. This intervention is not expected to significantly improve outcomes.
  Arms: Minimal Intervention

SUMMARY:
The transition from pediatric to adult IBD care can be stressful and wrought with challenges including access to care and establishment of new physician-patient relationships. There a few studies which characterize patterns of healthcare utilization during this critical period and its impact on outcomes. We hypothesize that uninterrupted healthcare utilization in academic centers and optimized communication with patients during the pediatric-adult transition period is associated with lower hospitalizations and surgery. This hypothesis will be addressed by a randomized clinical trial to determine the impact of monthly regular telephone contact with an IBD Registered Nurse versus standard of care during the pediatric-adult transition period. Outcomes will include healthcare utilization, health-related quality of life, patient satisfaction, and treatment adherence over 12 months of follow-up. Randomization and analyses will be stratified by whether subjects were transferred to adult care in an academic center or in a community practice. We hope that this research will facilitate optimal delivery of healthcare during the pediatric-adult transition.

DETAILED DESCRIPTION:
Rationale: The years marking the transition from pediatric-to-adult transition can be particularly difficult and transitioning patients with IBD may be at increased risk for loss to follow-up. As patient advocates, we need an intervention that would enable continuity of care especially among young adults who may face obstacles in accessing regular office visits. An intervention such as regular email contact with an IBD nurse may especially benefit those who are transitioning to community gastroenterology practices or to geographic regions where there is difficulty in accessing gastroenterology care. The lack of continuity of care may lead to delayed treatment which may be associated with poor clinical outcomes.

Research Question and Hypothesis: Our primary question is whether regular email contact with an IBD nurse can improve health outcomes. We hypothesize that such interaction, through augmented continuity of care will lead to increased patient satisfaction, increased medical adherence, improved transition readiness, decreased disease activity, and consequently decreased costly visits to the emergency department and hospitalizations.

Study Design: Multi-center randomized controlled clinical trial

Study population and inclusion/exclusion criteria: This study comprise adolescent subjects recruited from the IBD clinics of the Hospital for Sick Children, McMaster Children's Hospital or Children's Hospital of Eastern Ontario who meet the following inclusion criteria: (1) diagnosis of IBD; (2) at least age 16 years or older; (3) planning to undergo transition of care and will be followed by a gastroenterologist in either an academic center or the community; (4) have access to email or other means of telecommunication. We will exclude any subjects who will not be residing in Canada or who will not be enrolled in the Ontario Health Insurance Plan after exiting pediatric care. Registration with OHIP, even if residing in a different province, is required for monitoring of health utilization.

Health Implications: Our study may demonstrate cost-savings from decreased non-routine healthcare utilization coupled with improvement in health outcomes that may support the more widespread use of routine email-based interactions with IBD allied health providers in the pediatric-adult transition period.

ELIGIBILITY:
Inclusion Criteria:

* This study comprises adolescent subjects recruited from the IBD clinics of the Hospital for Sick Children and McMaster Children's Hospital who meet the following inclusion criteria: (1) diagnosis of IBD; (2) at least age 16 years or older; (3) planning to undergo transition of care and will be followed by a gastroenterologist in either an academic center or the community; (4) have access to email or other means of telecommunication.

Exclusion Criteria:

* We will exclude any subjects who will not be residing in Canada or who will not be enrolled in the Ontario Health Insurance Plan (OHIP) after exiting pediatric care. Registration with OHIP, even if residing in a different province, is required for the monitoring of health utilization.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2014-07; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Patient Satisfaction | Patient satisfaction will be assessed prior to transfer of care (within 3 months from the time of randomization) and again post-transfer of care (within 12 months from the time of randomization).
  A comprehensive study questionnaire containing the CACHE questionnaire will be administered to assess patient satisfaction.
  Reference: Casellas F, Ginard D, Vera I, Torrejón A. Development and testing of a new instrument to measure patient satisfaction with health care in inflammatory bowel disease: the CACHE questionnaire. Inflamm Bowel Dis. 2013 Mar;19(3):559-68.
Change in Medication Adherence | Medication adherence will be assessed prior to transfer of care (within 3 months from the time of randomization) and again post-transfer of care (within 12 months from the time of randomization).
  Medication adherence will be assessed with a comprehensive study questionnaire containing the Morisky questionnaire.
  Reference: Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care 1986;24:67-74.
Change in Non-Routine Healthcare Utilization | Non-routine healthcare utilization will be assessed retrospectively for 12 months prior to transfer of care and compared to 12 months post-transfer of care.
  IBD related clinic visits, admissions to hospital, emergency department visits, endoscopy and operative procedures, imaging procedures will all be recorded via telephone interview with the patient and also via linkage to the Institute of Clinical and Evaluative Sciences Databases which record health claims by Ontario residents . The date of transfer of care to an adult gastroenterologist will be recorded as well as any continuing appointments with a pediatric gastroenterologist beyond the transfer date.
Change in Transition Readiness | Transition readiness will be assessed prior to transfer of care (within 3 months from the time of randomization) and again post-transfer of care (within 12 months from the time of randomization).
  The Transition Readiness Assessment Questionnaire will be administered.
  Reference: Sawicki GS, Lukens-Bull K, Yin X, Demars N, Huang IC, Livingood W, Reiss J, Wood D. Measuring the transition readiness of youth with special healthcare needs: validation of the TRAQ--Transition Readiness Assessment Questionnaire. J Pediatr Psychol. 2011 Mar;36(2):160-71.

SECONDARY OUTCOMES:
Change in Quality of Life | Quality of life will be assessed prior to transfer of care (within 3 months from the time of randomization) and again post-transfer of care (within 12 months from the time of randomization).
  Health Related Quality of Life will be monitored by the Inflammatory Bowel Disease Questionnaire (IBDQ) validated in IBD patients.
  Reference: Inflammatory Bowel Disease Questionnaire - Guyatt G, Mitchell A, Irvine EJ, Singer J, Williams N, Goodacre R, Tompkins C. A new measure of health status for clinical trials in inflammatory bowel disease. Gastroenterology. 1989;96:804-10.
Change in Disease Activity | Disease activity will be assessed prior to transfer of care (within 3 months from the time of randomization) and again post-transfer of care (within 12 months from the time of randomization).
  Disease activity will be monitored using the Harvey Bradshaw Index (HBI) for Crohn's Disease related disease activity and the Ulcerative Colitis Disease Activity Index (UCDAI) for UC-related disease activity
  References:
  Harvey RF, Bradshaw JM. A simple index of Crohn's-disease activity. Lancet. 1980;315(8167):514.
  Sutherland LR, Martin F, Greer S, Robinson M, Greenberger N, Saibil F, Martin T, Sparr J, Prokipchuk E, Borgen L: 5-Aminosalicylic acid enema in the treatment of distal ulcerative colitis, proctosigmoiditis, and proctitis. Gastroenterology 1987, 92:1894-8.
Change in Knowledge of Disease | Knowledge of disease will be assessed prior to transfer of care (within 3 months from the time of randomization) and again post-transfer of care (within 12 months from the time of randomization).
  The Crohn's and Colitis Knowledge Questionnaire will be used to assess IBD specific knowledge.
  Reference: Eaden JA, Abram K, Mayberry JF. The Crohn's and colitis knowledge score: a test for measuring patient knowledge in inflammatory bowel disease. Am J Gastroenterol; 1999: 94(12):3560 - 3566.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Nguyen, MD, PhD, Principal Investigator — Mount Sinai Hospital, Canada; Anne Griffiths, MD, Principal Investigator — The Hospital For Sick Children, Toronto, Canada
Locations (3):
- Canada (3):
  - McMaster University Medical Center, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bollegala N, Brill H, Marshall JK. Resource utilization during pediatric to adult transfer of care in IBD. J Crohns Colitis. 2013 Mar;7(2):e55-60. doi: 10.1016/j.crohns.2012.05.010. Epub 2012 Jun 5. PMID 22677118
- [Background] Pinzon JL, Jacobson K, Reiss J. Say goodbye and say hello: the transition from pediatric to adult gastroenterology. Can J Gastroenterol. 2004 Dec;18(12):735-42. doi: 10.1155/2004/474232. PMID 15605138
- [Background] Baldassano R, Ferry G, Griffiths A, Mack D, Markowitz J, Winter H. Transition of the patient with inflammatory bowel disease from pediatric to adult care: recommendations of the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. J Pediatr Gastroenterol Nutr. 2002 Mar;34(3):245-8. doi: 10.1097/00005176-200203000-00001. No abstract available. PMID 11964946
- [Background] Scal P, Evans T, Blozis S, Okinow N, Blum R. Trends in transition from pediatric to adult health care services for young adults with chronic conditions. J Adolesc Health. 1999 Apr;24(4):259-64. doi: 10.1016/s1054-139x(98)00127-x. PMID 10227345
- [Background] Dabadie A, Troadec F, Heresbach D, Siproudhis L, Pagenault M, Bretagne JF. Transition of patients with inflammatory bowel disease from pediatric to adult care. Gastroenterol Clin Biol. 2008 May;32(5 Pt 1):451-9. doi: 10.1016/j.gcb.2008.01.044. Epub 2008 May 8. PMID 18472377
- [Background] Hait EJ, Barendse RM, Arnold JH, Valim C, Sands BE, Korzenik JR, Fishman LN. Transition of adolescents with inflammatory bowel disease from pediatric to adult care: a survey of adult gastroenterologists. J Pediatr Gastroenterol Nutr. 2009 Jan;48(1):61-5. doi: 10.1097/MPG.0b013e31816d71d8. PMID 19172125
- [Background] Greenley RN, Stephens M, Doughty A, Raboin T, Kugathasan S. Barriers to adherence among adolescents with inflammatory bowel disease. Inflamm Bowel Dis. 2010 Jan;16(1):36-41. doi: 10.1002/ibd.20988. PMID 19434722